CLINICAL TRIAL: NCT02486874
Title: Clinical Evaluation of PoreSkin: A Human Acellular Dermal Matrix
Brief Title: Clinical Evaluation of PoreSkin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Apichai Angspatt, Apichai Angspatt, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 283/52
Record Dates: First submitted 2015-06-03; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-05

CONDITIONS: Treatment
Keywords: Human acellular dermal matrix, burns, wound healing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): PoreSkin, a human acellular dermal matrix, were used for scar contracture treatment
  Interventions: Device: PoreSkin

INTERVENTIONS:
Device: PoreSkin — a human acellular dermal matrix

SUMMARY:
PoreSkin, a human acellular dermal matrix (hADM) manufactured by Faculty of Medicine, Chulalongkorn University, is the first human dermal substitute developed in Thailand. It is a permanent dermal substitute aiming to reduce skin contracture. The objective of this study is to assess the safety and ability in achieving durable and cosmetic coverage of PoreSkin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 18-60 years with burn scar contracture and hypertrophic scar

Exclusion Criteria:

* Undergoing immunosuppressive therapy
* Immunocompromise host (DM, HIV infected)
* Evidence of malnutrition
* Active malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The engraftment rate | 1 month

SECONDARY OUTCOMES:
Any local complications | 1 month
  erythema, infection, fever, and rejection of the graft
the final cosmetic result | 1 month
  evaluated by Vancouver Scar scale